CLINICAL TRIAL: NCT01849874
Title: The MILO Study (MEK Inhibitor in Low-grade Serous Ovarian Cancer): A Multinational, Randomized, Open-label Phase 3 Study of MEK162 vs. Physician's Choice Chemotherapy in Patients With Recurrent or Persistent Low-grade Serous Carcinomas of the Ovary, Fallopian Tube or Primary Peritoneum
Brief Title: A Study of MEK162 vs. Physician's Choice Chemotherapy in Patients With Low-grade Serous Ovarian, Fallopian Tube or Peritoneal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per recommendation of the DMC, enrollment into the study was discontinued in April 2016 after the planned interim efficacy analysis showed the hazard ratio for PFS crossed the predefined futility boundary.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-162-311; C4211003 (Other: Alias Study Number); 2013-000277-72 (EudraCT Number)
Record Dates: First submitted 2013-05-06; First posted 2013-05-09 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Low-grade Serous Ovarian Cancer; Low-grade Serous Fallopian Tube Cancer; Low-grade Serous Peritoneal Cancer
MeSH Terms: interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEK162 (Experimental)
  Interventions: Drug: MEK162, MEK inhibitor; oral
- Physician's choice chemotherapy (Active Comparator)
  Interventions: Drug: Physician's choice chemotherapy

INTERVENTIONS:
Drug: MEK162, MEK inhibitor; oral — multiple dose, single schedule
  Arms: MEK162
Drug: Physician's choice chemotherapy — Patients will receive one of the following chemotherapies as determined by the physician:
  * Liposomal doxorubicin, anthracycline antibiotic; intravenous (multiple dose, single schedule)
  * Paclitaxel, mitotic inhibitor; intravenous (multiple dose, single schedule)
  * Topotecan, topoisomerase 1 inhibitor; intravenous (multiple dose, single schedule)
  Arms: Physician's choice chemotherapy

SUMMARY:
The MILO Study (MEK Inhibitor in Low-grade Serous Ovarian Cancer) is a Phase 3 study during which patients with recurrent or persistent low-grade serous (LGS) carcinomas of the ovary, fallopian tube or primary peritoneum will receive either investigational study drug MEK162 or a chemotherapy chosen by the physician (liposomal doxorubicin, paclitaxel or topotecan). Patients will be followed to compare the effectiveness of the study drug to that of the selected chemotherapies. Patients may be eligible to crossover from physician's choice chemotherapy to MEK162 if they meet certain inclusion criteria including centrally confirmed disease progression. Approximately 360 patients from North America, Europe and Australia will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of LGS carcinoma of the ovary, fallopian tube or primary peritoneum (invasive micropapillary serous carcinoma or invasive grade 1 serous carcinoma), confirmed histologically and verified by central pathology review.
* Recurrent or persistent measurable disease that has progressed (defined as radiological and/or clinical progression; an increase in cancer antigen [CA]-125 alone is not sufficient) on or after last therapy (i.e., chemotherapy, hormonal therapy, surgery) and is not amenable to potentially curative intent surgery, as determined by the patient's treating physician.
* Must have received at least 1 prior platinum-based chemotherapy regimen but have received no more than 3 lines of prior chemotherapy regimens, with no limit to the number of lines of prior hormonal therapy. Front-line therapy may include neoadjuvant and adjuvant therapy and will be counted as 1 prior systemic regimen. Biological therapy (e.g. bevacizumab) administered as a single agent is considered a prior systemic regimen and not a prior chemotherapy regimen. Maintenance therapy is not considered its own regimen but should be included with the regimen that it follows.
* Available archival tumor sample (excisional or core biopsy) for confirmation of LGS carcinoma diagnosis. If adequate archival tumor sample is not available, willingness to consent to tissue biopsy.
* Suitable for treatment with at least one of the physician's choice chemotherapy options (liposomal doxorubicin, paclitaxel or topotecan) as determined by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Additional criteria exist.

Key Exclusion Criteria:

* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).
* Prior therapy with a MEK or BRAF inhibitor.
* History of Gilbert's syndrome.
* Impaired cardiovascular function or clinically significant cardiovascular diseases.
* Uncontrolled or symptomatic brain metastases that are not stable or require steroids, are potentially life-threatening or have required radiation within 28 days prior to first dose of study treatment.
* Concomitant malignancies or previous malignancies with less than a 5-year disease-free interval at the time of first dose of study treatment; patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or ductal carcinoma in situ may be enrolled irrespective of the time of diagnosis.
* Known positive serology for the human immunodeficiency virus (HIV), active hepatitis B and/or active hepatitis C.
* Prior randomization into this clinical study.
* Additional criteria exist.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 341 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (224):
- United States (77):
  - University of Arizona Cancer Center, Phoenix, Arizona
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - Oncology Research Associates, PLLC d/b/a Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Keck Hospital of USC, Los Angeles, California
  - LAC & USC Medical Center, Los Angeles, California
  - USC Healthcare Consultation Center 1, Los Angeles, California
  - USC Healthcare Consultation Center 2, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Admin.Office/Study Supplies Mailing Address: UCLA Medicine Hematology-Oncology, Los Angeles, California
  - Doris Stein Research Center Building, Los Angeles, California
  - University of California Los Angeles, Hematology-Oncology Clinic, Los Angeles, California
  - Gynecologic Oncology Associates, Newport Beach, California
  - University of California, Irvine/UC Irvine Health, Orange, California
  - UCLA Hematology/Oncology Clinic - Santa Monica, Santa Monica, California
  - UCLA Hematology Oncology Clinic Santa Clarita, Valencia, California
  - UCLA Hematology - Oncology Clinic - Westlake Village, Westlake Village, California
  - Rocky Mountain Lions Eye Institute, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Colorado Denver, University of Colorado Cancer Center, Aurora, Colorado
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Eye Physicians of Central Florida, Maitland, Florida
  - Florida Hospital, Orlando, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Eye Physicians of Central, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Florida Cancer Specialists, Wellington, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Georgia Regents University Cancer Center, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - St. Vincent Cancer Care, Indianapolis, Indiana
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - St. Vincent Gynecology Oncology, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Inc., Indianapolis, Indiana
  - Associated Vitreoretinal and Uveitis Consultants, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston (OCB), Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Kresge Eye Institute, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Center For Clinical Studies, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center - Einstein Center for Cancer Care, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Montefiore Medical Center - Centennial Women's Health, The Bronx, New York
  - Montefiore Medical Center, Green Medical Arts Pavilion, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Fairview Hospital Moll Pavilion Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cleveland Clinic-Main Campus, Cleveland, Ohio
  - James Cancer Hospital & Solove Research Institute, Columbus, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Stefanie Spielman Comprehensive Breast Cancer, Columbus, Ohio
  - OSU Gynecologic Oncology at Mill Run, Hilliard, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - University of Cincinnati Physicians Company, West Chester, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Stephenson Cancer Center(clinic location), Oklahoma City, Oklahoma
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jeanes Hospital, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Parkland Health and Hospital System, Dallas, Texas
  - UT Southwestern Medical Center-Zale Lipshy University Hospital, Dallas, Texas
  - UT Southwestern Medical Center-Clements University Hospital, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Australia (11):
  - Dr Anil Arora, Wahroonga, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Mater Misericordiae Health Services Brisbane Limited, South Brisbane, Queensland
  - Adelaide Cardiology, Adelaide, South Australia
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Thomas and Delaney Optometrists, Norwood, South Australia
  - Burnside War Memorial Hospital, Toorak Gardens, South Australia
  - Sunshine Hospital, St Albans, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Innsbruck Medical University, Innsbruck, Tyrol, Austria
- Belgium (9):
  - Centre Hospitalier de l'ardenne, Libramont, Luxembourg
  - Private practice Ophthalmology, Libramont, Luxembourg
  - University Hospital Leuven, Leuven, Vlaams-brabant
  - Cliniques Universitaires Saint-Luc, Brussels
  - Ghent University Hospital, Ghent
  - University Hospital Gent, Ghent
  - CHR de la Citadelle, Liège
  - Clinique et Maternite Sainte-Elisabeth Namur, Namur
  - Sint-Augustinus, Wilrijk
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Center, Department of Oncology, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (Chum) - Hopital Notre-Dame, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Czechia (6):
  - Teaching Hospital Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - General University Hospital in Prague, Prague
- Denmark (7):
  - Aalborg Sygehus Apotek, Aalborg, North Jutland
  - Aalborg University Hospital, Aalborg, North Jutland
  - Herlev Hospital Onkologisk AFD, Herlev
  - Ojenklinikken 2061, København Ø
  - Radiologisk Afdeling 2023, København Ø
  - Region Hovedstadens Apotek, København Ø
  - Rigshospitalet, København Ø
- Tampere University Hospital, Tampere, Finland
- France (17):
  - CHU Jean Minjoz, Besançon
  - Centre Oscar Lambret, Lille
  - Hopital Prive La Louviere, Lille
  - Hopital Edouard Herriot, Lyon
  - Centre Leon Berard, Lyon
  - Centre Paradis Monticelli, Marseille
  - Institut Paoli Calmettes - Departement d'Oncologie Medicale, Marseille
  - Centre d'Ophtalmologie du LEZ Centre Medical Les Roques, Montferrier S/lez
  - Institut Regional du Cancer Montpellier, Montpellier
  - Cabinet Liberal du Dr Xavier Zanlonghi, Nantes
  - Clinique Sourdille, Nantes
  - L'Hopital Prive du Confluent SAS, Nantes
  - Centre d'Investigations Cliniques 1423, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Investigateur CARIO - HPCA, Plérin
  - Institut de Cancerologie de I'Ouest - Rene Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Germany (12):
  - Universitaets-Brustzentrum, Tübingen, Baden-Wurttemberg
  - Universitätsfrauenklinik Ulm, Ulm, Baden-Wurttemberg
  - Klinikum rechts der Isar, Munich, Bavaria
  - Klinik fur Frauenheilkunde und Geburtshilfe, Kassel, Hesse
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - Uni Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Charité Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinik Freiburg, Freiburg im Breisgau
  - Frauenheilkunde und Geburtshilfe, Greifswald
  - NCT Nationales Centrum für Tumorerkrankungen Heidelberg, Heidelberg
- Hungary (9):
  - Euromedic Diagnostics Magyarorszag Kft., Győr, Győr-Moson-Sopron
  - Petz Aladar Korhaz Kardiologiai Osztaly, Győr, Győr-Moson-Sopron
  - Petz Aladar Korhaz Szemeszeti Osztaly, Győr, Győr-Moson-Sopron
  - Magyar Honvedseg Egeszsegugyi Kozpont, Onkologiai Osztaly, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem AOK Szemeszeti Klinika, Budapest
  - Orszagos Onkologiai Intezet Kozponti Aneszteziologiai es Intenzivterapias Osztaly, Budapest
  - Orszagos Onkologiai Intezet, Nogyogyaszati Osztaly, Budapest
  - Orszagos Onkologiai Intezet, Budapest
- St James's Hospital, Dublin, Dublin 8, Ireland
- Italy (26):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Centro di Riferimento Oncologico - Struttura Operativa Complessa (SOC)- Oncologia Medica C, Aviano, Pordenone
  - Ospedale Civile degli Infermi - Servizio di Oculistica, Faenza, Ravenna
  - Ospedale Civile degli Infermi - Unita Operativa di Oncologia Medica, Faenza, Ravenna
  - Ospedale Umberto I - Unita Operativa di Oncologia, Lugo, Ravenna
  - Istituto Nazionale Tumori Regina Elena - Oncologia Medica A, Roma, RM
  - Policlinico Umberto I - Università Sapienza, Roma, ROME
  - Azienda Ospedaliera Sant' Andrea - Unita Operativa Semplice di Patologia Vitreo-Retinica, Roma, ROME
  - SSD Oncologia Medica Addarii-Zamagni - Policlinico S. Orsola-Malpighi, Bologna
  - Struttura Complessa di Oftalmologia Policlinico S. Orsola-Malpighi, Bologna
  - Spedali Civili di Brescia - Struttura Complessa Clinicizzata - U.O.di Oculistica, Brescia
  - Spedali Civili Di Brescia, Brescia
  - Azienda Ospedaliera Cannizzaro, Catania
  - Ospedale San Raffaele - Unita Operativa di Oculistica, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori - SC Oncologia Ginecologica, Milan
  - Istituto Europeo Oncologico, Milan
  - Azienda Ospedaliera Vincenzo Monaldi di Napoli - U.O.C. di Oculistica, Napoli
  - Istituto Nazionale Tumori di Napoli, "G.Pascale" , Oncologia Medica, Dipartimento Uro-Ginecologico, Napoli
  - Universita degli Studi Federico II di Napoli Dipartimento di Neuroscienze Scienze, Napoli
  - Universita degli Studi Federico II di Napoli Oncologia Medica, Napoli
  - Azienda Opsedaliera S. Maria Degli Angeli Pordenone-Dipartimento di Chirurgia Specialistica -, Pordenone
  - Ospedale Santa Maria delle Croci - Oculistica, Ravenna
  - Ospedale Santa Maria delle Croci - Unita Operativa di Oncologia, Ravenna
  - Dipartimento Organi di Senso, Roma
  - Dipartimento di Scienze Chirurgiche per le Patologie della Testa e del Collo - UOC di Oculistica, Roma
  - Policlinico Agostino Gemelli, Roma
- Netherlands (3):
  - Academic Medical Center (AMC), Amsterdam, North Holland
  - University Medical Center Groningen, Medical Oncology, Groningen
  - Maastricht University Medical Centre, Maastricht
- Norway (3):
  - Aleris, Oslo
  - Avd. for gynekologisk kreft, Radiumhospitalet, Oslo
  - Oslo Universitetssykehus HF, Oslo
- Centralny Szpital Kliniczny MON, Warsaw, Poland
- Spain (19):
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Reina Sofía/ Provincial, Córdoba, Castille-La Mancha
  - Centro de Salud Anoeta, Anoeta, Guipuzcoa
  - Hospital Universitario Donostia, Donostia / San Sebastian, Guipuzcoa
  - Ophthalmology at Instituto Oftalmologico Integral, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de Sant Joan Despi Moises Broggi, Barcelona
  - Cardiology at Consulta de Cardiologia, Córdoba
  - Centro Medico Sanitas Ressalta, Córdoba
  - Instituto de Oftalmologia y Hospital La Arruzafa, Córdoba
  - Radiology at Centro Medico Sanitas Ressalta, Córdoba
  - Radiology at Hospital Univeristari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen de la Salud, Toledo
  - Fundacion IVO-Instituto Valenciano de Oncologia, Valencia
  - Ophthalmology at Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (2):
  - Karolinska Universitetssjukhuset, Stockholm
  - Onkologkliniken Akademiska Sjukhuset, Uppsala
- United Kingdom (12):
  - Sarah Cannon Research Institute UK, London, England
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - University of Nottingham, Nottingham, Nottinghamshire
  - Ashtead Hospital, Ashtead, Surrey
  - The Clock House Medical Practice, Epsom, Surrey
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - St. Anthony's Hospital, North Cheam, Sutton
  - City Hospital, Birmingham, WEST Midlands
  - Royal Marsden NHS Foundation Trust, London
  - The Harley Street Clinic, London
  - London Eye Diagnostic Centre, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Grisham RN, Vergote I, Banerjee S, Drill E, Kalbacher E, Mirza MR, Romero I, Vuylsteke P, Coleman RL, Hilpert F, Oza AM, Westermann A, Oehler MK, Pignata S, Aghajanian C, Colombo N, Cibula D, Moore KN, Del Campo JM, Berger R, Marth C, Sehouli J, O'Malley DM, Churruca C, Kristensen G, Clamp A, Farley J, Iyer G, Ray-Coquard I, Monk BJ. Molecular Results and Potential Biomarkers Identified from the Phase 3 MILO/ENGOT-ov11 Study of Binimetinib versus Physician Choice of Chemotherapy in Recurrent Low-Grade Serous Ovarian Cancer. Clin Cancer Res. 2023 Oct 13;29(20):4068-4075. doi: 10.1158/1078-0432.CCR-23-0621. PMID 37581616
- [Derived] Monk BJ, Grisham RN, Banerjee S, Kalbacher E, Mirza MR, Romero I, Vuylsteke P, Coleman RL, Hilpert F, Oza AM, Westermann A, Oehler MK, Pignata S, Aghajanian C, Colombo N, Drill E, Cibula D, Moore KN, Christy-Bittel J, Del Campo JM, Berger R, Marth C, Sehouli J, O'Malley DM, Churruca C, Boyd AP, Kristensen G, Clamp A, Ray-Coquard I, Vergote I. MILO/ENGOT-ov11: Binimetinib Versus Physician's Choice Chemotherapy in Recurrent or Persistent Low-Grade Serous Carcinomas of the Ovary, Fallopian Tube, or Primary Peritoneum. J Clin Oncol. 2020 Nov 10;38(32):3753-3762. doi: 10.1200/JCO.20.01164. Epub 2020 Aug 21. PMID 32822286

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As of the data cutoff date of 20 Jan 2016 for primary completion date (PCD), a total of 303 participants were enrolled, with 201 (200 treated) in MEK162 group and 102 (94 treated) in physician's choice group. After PCD, additional 27 participants were enrolled in MEK162 group and 11 in physician's choice group. Data reported was based on the last participant last visit date (23 Aug 2022). Note: one participant was enrolled before PCD and received the first dose after PCD.
Groups:
- MEK162: Participants received an oral dose of 45 milligram (mg) of MEK162 tablets (3 tablets of 15 mg) twice daily for each 28-day treatment cycle until disease progression, withdrawal of consent, initiation of subsequent anticancer therapy, lost to follow-up or death, whichever occurred first. Participants were followed up to 30 days after last dose of study intervention.
- Physician's Choice: Participants received chemotherapies as per treating physician's choice in accordance to the institutional standard of care. Participants received one of the three intravenous (IV) infusion therapies: Liposomal doxorubicin 40 milligram per meter square (mg/m^2) on Day 1 of each 28-day cycle or Paclitaxel 80 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle or, Topotecan 1.25 mg/m^2 on Days 1 through 5 of each 21-day cycle. Participants were followed up to 30 days after last dose of study intervention.
Period: Overall Study
Arm/Group | MEK162 | Physician's Choice
Started | 228 | 113
Treated | 227 | 106
Safety Population (Safety population consisted of all participants who received at any dose of study intervention (MEK162 or physician's choice chemotherapy).) | 227 (The safety population number reported as "At risk" in AE section.) | 106 (The safety population number reported as "At risk" in AE section.)
Crossover Period (After failure of physician's choice chemotherapy in the randomized period, participants entered into the crossover period to receive MEK162 treatment 45 mg orally twice daily with water irrespective of food, continuously, starting on Day 1 of the crossover period. Crossover from physician's choice chemotherapy treatment to MEK162 treatment was no longer permitted after enrollment was early discontinued.) | 0 | 18 (No data, safety or efficacy, were collected for crossover set, as the crossover period was stopped early.)
Completed | 0 | 0
Not Completed | 228 | 113
Not completed — Death | 89 | 42
Not completed — Withdrawal by Subject | 17 | 16
Not completed — Lost to Follow-up | 3 | 2
Not completed — Study Termination By Sponsor | 93 | 48
Not completed — Completed as per protocol amendment 6 | 3 | 0
Not completed — Physician Decision | 7 | 1
Not completed — Other | 16 | 4

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants in the safety population. Safety population consisted of all participants who received at any dose of study intervention (MEK162 or physician's choice chemotherapy).
Groups:
- Total: Total of all reporting groups
Arm/Group | MEK162 | Physician's Choice | Total
Number analyzed (Participants) | 227 | 106 | 333
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.26 (14.64) | 50.12 (13.35) | 51.58 (14.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227 | 106 | 333
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 9 | 27
  Not Hispanic or Latino | 200 | 95 | 295
  Unknown or Not Reported | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the earliest documented disease progression date or death due to any cause whichever occurred first. Disease progression was defined as at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including Baseline) and an absolute increase of greater than or equal to (>=) 5 millimeter (mm). Appearance of new lesions >=10 mm in diameter also constituted PD. If a participant did not have an event at the time of the analysis cutoff or at the start of any new therapy, PFS was censored at the date of last adequate tumor assessment.
Time Frame: From randomization until documented progressive disease (PD) or death, whichever occurred first, for censored participants at the date of last adequate tumor assessment (up to 24 months)
Population: Analysis population included all randomized participants as of PCD (201 participants in MEK162 group and 102 participants in physician's choice group). In the futility analysis based on PCD, the futility boundary was crossed, and therefore, no additional efficacy data was collected due to study early termination and no additional efficacy analyses were conducted.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MEK162 | Physician's Choice
Number analyzed (Participants) | 201 | 102
months | 9.10 [7.29 to 11.30] | 10.58 [9.20 to 14.52]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants who were alive at the data cutoff date were censored for overall survival at their last contact date.
Time Frame: From randomization date to the date of death, for censored participants at their last contact date (up to 24 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MEK162 | Physician's Choice
Number analyzed (Participants) | 201 | 102
months | 25.33 [18.46 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 20.83 [17.45 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events.

3. Secondary Outcome: Objective Response Rate Per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (RECIST V1.1)
Description: ORR was defined as the percentage of participants achieving an overall best response of complete response (CR) or partial response (PR) (responders). CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures less than (<) 10 mm, PR was defined as at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the Baseline sum of diameters. Non-target lesions must be non-progressive disease.
Time Frame: From randomization until disease progression or death (up to 24 months)
Population: Analysis population included all randomized participants with measurable disease at baseline per BICR as of PCD (198 participants in MEK162 group and 101 participants in physician's choice group). In the futility analysis based on PCD, the futility boundary was crossed, and therefore, no additional efficacy data was collected due to study early termination and no additional efficacy analyses were conducted.
Measure: Number; unit: percentage of participants
Arm/Group | MEK162 | Physician's Choice
Number analyzed (Participants) | 198 | 101
percentage of participants | 16 | 13

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from first radiographic evidence of response to the earliest documented progression date or death due to any cause, and was calculated on responders only. Responders with no PD or death date or subsequent anticancer therapy by the data cutoff date, were censored for DOR at their last radiological assessment. Responders who received subsequent anticancer therapy prior to PD or death were censored at their last radiological assessment prior to initiation of subsequent anticancer therapy.
Time Frame: From the first radiographic evidence of response to the first documentation of PD or death, for censored participants at their last radiological assessment (up to 24 months)
Population: Analysis population included all randomized participants with measurable disease at baseline per BICR with response ongoing as of PCD (23 in MEK162 group and 8 in physician's choice group). Here, "Number of Participants Analyzed" signifies number of participants evaluable for DOR. In the futility analysis based on PCD, the futility boundary was crossed, and therefore, no additional efficacy data was collected due to study early termination and no additional efficacy analyses were conducted.
Measure: Median (Full Range); unit: months
Arm/Group | MEK162 | Physician's Choice
Number analyzed (Participants) | 23 | 8
months | 8.05 [0.03 to 11.99] | 6.67 [0.03 to 9.69]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate was defined as percentage of participants with disease control. Disease control was defined as a best response of CR or PR, or stable disease (SD) documented at Week 24 or later. CR was defined as disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm, and PR is defined as at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the Baseline sum of diameters. Non-target lesions must be non-progressive disease. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters on study.
Time Frame: Week 24
Population: Due to the lack of follow-up data as of PCD, data for this outcome measure was not collected. In the futility analysis based on PCD, the futility boundary was crossed, and therefore, no additional efficacy data was collected due to study early termination and no additional efficacy analyses were conducted.
Arm/Group | MEK162 | Physician's Choice
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From the first dose of study intervention until 30 days after the last dose (up to 9 years)
Population: The safety set included all participants who received at least 1 dose of study intervention and had at least 1 post-treatment assessment, including death. No data was collected for the crossover set due to the early stopping of the crossover period.
Measure: Count of Participants; unit: Participants
Arm/Group | MEK162 | Physician's Choice
Number analyzed (Participants) | 227 | 106
Participants
  AEs | 227 | 105
  SAEs | 126 | 31

7. Secondary Outcome: Number of Participants With Shift Greater Than or Equal to Grade 3 From Baseline in Laboratory Parameter Values Based on National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03
Description: Number of participants with shifts from normal Baseline values (Grade 0) to abnormal post-baseline values on-study (shift to greater than or equal to Grade 3) were reported as per NCI-CTCAE, v4.03 graded from Grade 1 to 5. Grade 1: Mild; asymptomatic/ mild symptoms; clinical/diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local/noninvasive intervention indicated. Grade 3: Severe/medically significant but not immediately life-threatening; hospitalization/prolongation of hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death. Shifts in lab parameter from Grade 0 to 3, Grade 0 to 4 and Grade 0 to Low 3 and 4 and Grade 0 to High 3 and 4 (for parameters total hemoglobin, lymphocytes, white blood cells, calcium, magnesium, potassium, and sodium) were reported.
Time Frame: From the first dose of study intervention until 30 days after the last dose (up to 9 years)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | MEK162 | Physician's Choice
Number analyzed (Participants) | 227 | 106
Participants
  International Normalized Ratio: Grade 0 to 3 | 0 | 0
  International Normalized Ratio: Grade 0 to 4 | 0 | 0
  Neutrophils: Grade 0 to 3 | 3 | 7
  Neutrophils: Grade 0 to 4 | 0 | 1
  Platelet Count: Grade 0 to 3 | 0 | 0
  Platelet Count: Grade 0 to 4 | 1 | 0
  Partial Thromboplastin Time: Grade 0 to 3 | 4 | 2
  Partial Thromboplastin Time: Grade 0 to 4 | 0 | 0
  Total Hemoglobin: Grade 0 to Low 3 | 10 | 2
  Total Hemoglobin: Grade 0 to Low 4 | 0 | 0
  Total Hemoglobin: Grade 0 to High 3 | 0 | 0
  Total Hemoglobin: Grade 0 to High 4 | 0 | 0
  Lymphocytes: Grade 0 to Low 3 | 8 | 3
  Lymphocytes: Grade 0 to Low 4 | 1 | 0
  Lymphocytes: Grade 0 to High 3 | 0 | 0
  Lymphocytes: Grade 0 to High 4 | 0 | 0
  White Blood Cells: Grade 0 to Low 3 | 0 | 1
  White Blood Cells: Grade 0 to Low 4 | 0 | 1
  White Blood Cells: Grade 0 to High 3 | 0 | 0
  White Blood Cells: Grade 0 to High 4 | 0 | 0
  Albumin: Grade 0 to 3 | 1 | 1
  Albumin: Grade 0 to 4 | 0 | 0
  Alkaline Phosphatase: Grade 0 to 3 | 4 | 1
  Alkaline Phosphatase: Grade 0 to 4 | 0 | 0
  Alanine Aminotransferase/Serum Glutamic-Pyruvic Transaminase: Grade 0 to 3 | 7 | 1
  Alanine Aminotransferase/Serum Glutamic-Pyruvic Transaminase: Grade 0 to 4 | 0 | 0
  Aspartate Aminotransferase/Serum Glutamic-Oxaloacetic Transaminase: Grade 0 to 3 | 7 | 1
  Aspartate Aminotransferase/Serum Glutamic-Oxaloacetic Transaminase: Grade 0 to 4 | 0 | 0
  Creatine Kinase: Grade 0 to 3 | 52 | 0
  Creatine Kinase: Grade 0 to 4 | 12 | 0
  Serum Creatinine: Grade 0 to 3 | 1 | 0
  Serum Creatinine: Grade 0 to 4 | 0 | 0
  Total Bilirubin: Grade 0 to 3 | 1 | 0
  Total Bilirubin: Grade 0 to 4 | 0 | 0
  Calcium: Grade 0 to Low 3 | 0 | 1
  Calcium: Grade 0 to Low 4 | 1 | 1
  Calcium: Grade 0 to High 3 | 1 | 0
  Calcium: Grade 0 to High 4 | 0 | 0
  Magnesium: Grade 0 to Low 3 | 2 | 1
  Magnesium: Grade 0 to Low 4 | 0 | 0
  Magnesium: Grade 0 to High 3 | 1 | 0
  Magnesium: Grade 0 to High 4 | 0 | 0
  Potassium: Grade 0 to Low 3 | 10 | 4
  Potassium: Grade 0 to Low 4 | 0 | 0
  Potassium: Grade 0 to High 3 | 3 | 2
  Potassium: Grade 0 to High 4 | 0 | 0
  Sodium: Grade 0 to Low 3 | 5 | 2
  Sodium: Grade 0 to Low 4 | 1 | 0
  Sodium: Grade 0 to High 3 | 3 | 0
  Sodium: Grade 0 to High 4 | 1 | 0

8. Secondary Outcome: Quality of Life Per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 (QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item cancer-specific instrument that assesses participant reported outcomes, consisting of 5 functional scales, 3 symptoms scales, a global health status/quality of life (QOL) scale, and 6 single-item scales. The global health status/QOL scale has 7 possible scores of responses (1=very poor to 7=excellent). All other items have 4 possible scores (1=not at all, 2=a little, 3=quite a bit, 4=very much). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100, with 0 being the worst and 100 being the best for global health status/QOL and functional scales, and 0 being the best and 100 being the worst for symptoms scales. In this study, global health status/QOL scale score was identified as the primary patient-reported outcome variable of interest. Physical functioning, emotional functioning, and social functioning scale scores were considered as secondary. Higher scores indicate better quality of life.
Time Frame: Screening, every 8 weeks from randomization for the first 72 weeks (while on treatment), treatment discontinuation visit, 30-day safety follow-up visit
Population: Analysis population included all randomized participants (228 participants in MEK162 group, 113 participants in physician's choice group).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- MEK 162: Participants received an oral dose of 45 milligram (mg) of MEK162 tablets (3 tablets of 15 mg) twice daily for each 28-day treatment cycle until disease progression, withdrawal of consent, initiation of subsequent anticancer therapy, lost to follow-up or death, whichever occurred first. Participants were followed up to 30 days after last dose of study intervention.
Arm/Group | MEK 162 | Physician's Choice
Number analyzed (Participants) | 228 | 113
Scores on a scale
  Global health status/QOL Score at Screening: number analyzed (Participants) | 224 | 111
  Global health status/QOL Score at Screening | 67.2 (19.9) | 66.4 (24.5)
  Global health status/QOL Score at Week 9: number analyzed (Participants) | 180 | 82
  Global health status/QOL Score at Week 9 | 57.4 (19.4) | 66.4 (20.4)
  Global health status/QOL Score at Week 17: number analyzed (Participants) | 135 | 68
  Global health status/QOL Score at Week 17 | 58.4 (19.9) | 65.4 (17.5)
  Global health status/QOL Score at Week 25: number analyzed (Participants) | 108 | 47
  Global health status/QOL Score at Week 25 | 60.5 (18.7) | 65.4 (19.6)
  Global health status/QOL Score at Week 33: number analyzed (Participants) | 86 | 31
  Global health status/QOL Score at Week 33 | 60.4 (20.0) | 63.7 (18.9)
  Global health status/QOL Score at Week 41: number analyzed (Participants) | 77 | 25
  Global health status/QOL Score at Week 41 | 60.4 (18.6) | 73.0 (18.5)
  Global health status/QOL Score at Week 49: number analyzed (Participants) | 65 | 18
  Global health status/QOL Score at Week 49 | 60.9 (19.4) | 69.9 (17.9)
  Global health status/QOL Score at Week 57: number analyzed (Participants) | 43 | 16
  Global health status/QOL Score at Week 57 | 62.4 (18.3) | 76.6 (20.9)
  Global health status/QOL Score at Week 65: number analyzed (Participants) | 40 | 11
  Global health status/QOL Score at Week 65 | 60.8 (18.9) | 65.9 (22.8)
  Global health status/QOL Score at Week 73: number analyzed (Participants) | 34 | 8
  Global health status/QOL Score at Week 73 | 62.0 (19.7) | 67.7 (21.6)
  Global health status/QOL Score at Treatment Discontinuation Visit: number analyzed (Participants) | 114 | 46
  Global health status/QOL Score at Treatment Discontinuation Visit | 47.0 (21.4) | 60.9 (25.6)
  Global health status/QOL Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Global health status/QOL Score at 30-Day Safety Follow-up | 59.8 (19.1) | 69.3 (18.0)
  Physical functioning Score at Screening: number analyzed (Participants) | 225 | 111
  Physical functioning Score at Screening | 80.2 (19.2) | 82.6 (18.7)
  Physical functioning Score at Week 9: number analyzed (Participants) | 180 | 83
  Physical functioning Score at Week 9 | 74.8 (20.3) | 81.4 (18.4)
  Physical functioning Score at Week 17: number analyzed (Participants) | 138 | 68
  Physical functioning Score at Week 17 | 75.3 (19.5) | 79.4 (20.9)
  Physical functioning Score at Week 25: number analyzed (Participants) | 109 | 47
  Physical functioning Score at Week 25 | 75.5 (20.8) | 80.2 (19.9)
  Physical functioning Score at Week 33: number analyzed (Participants) | 86 | 31
  Physical functioning Score at Week 33 | 76.6 (19.6) | 81.5 (23.3)
  Physical functioning Score at Week 41: number analyzed (Participants) | 77 | 25
  Physical functioning Score at Week 41 | 75.1 (19.9) | 83.7 (21.9)
  Physical functioning Score at Week 49: number analyzed (Participants) | 65 | 18
  Physical functioning Score at Week 49 | 77.5 (18.0) | 83.7 (20.5)
  Physical functioning Score at Week 57: number analyzed (Participants) | 44 | 16
  Physical functioning Score at Week 57 | 74.8 (19.4) | 83.3 (20.7)
  Physical functioning Score at Week 65: number analyzed (Participants) | 41 | 11
  Physical functioning Score at Week 65 | 77.2 (19.7) | 81.8 (20.2)
  Physical functioning Score at Week 73: number analyzed (Participants) | 34 | 8
  Physical functioning Score at Week 73 | 77.2 (21.1) | 78.3 (25.6)
  Physical functioning Score at Treatment Discontinuation Visit: number analyzed (Participants) | 114 | 46
  Physical functioning Score at Treatment Discontinuation Visit | 66.6 (23.8) | 71.0 (25.0)
  Physical functioning Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Physical functioning Score at 30-Day Safety Follow-up | 71.7 (21.5) | 78.6 (23.4)
  Emotional functioning Score at Screening: number analyzed (Participants) | 225 | 111
  Emotional functioning Score at Screening | 75.8 (21.2) | 71.7 (24.0)
  Emotional functioning Score at Week 9: number analyzed (Participants) | 180 | 82
  Emotional functioning Score at Week 9 | 73.1 (21.6) | 75.8 (22.9)
  Emotional functioning Score at Week 17: number analyzed (Participants) | 136 | 68
  Emotional functioning Score at Week 17 | 73.9 (20.2) | 77.7 (19.1)
  Emotional functioning Score at Week 25: number analyzed (Participants) | 109 | 47
  Emotional functioning Score at Week 25 | 76.7 (20.0) | 78.7 (20.9)
  Emotional functioning Score at Week 33: number analyzed (Participants) | 86 | 31
  Emotional functioning Score at Week 33 | 75.1 (21.6) | 81.6 (20.4)
  Emotional functioning Score at Week 41: number analyzed (Participants) | 77 | 25
  Emotional functioning Score at Week 41 | 74.7 (22.0) | 79.0 (24.9)
  Emotional functioning Score at Week 49: number analyzed (Participants) | 65 | 18
  Emotional functioning Score at Week 49 | 77.6 (18.6) | 79.2 (24.0)
  Emotional functioning Score at Week 57: number analyzed (Participants) | 43 | 16
  Emotional functioning Score at Week 57 | 77.7 (18.7) | 81.8 (26.6)
  Emotional functioning Score at Week 65: number analyzed (Participants) | 40 | 11
  Emotional functioning Score at Week 65 | 77.1 (17.6) | 80.3 (28.7)
  Emotional functioning Score at Week 73: number analyzed (Participants) | 34 | 8
  Emotional functioning Score at Week 73 | 73.4 (22.5) | 69.8 (31.5)
  Emotional functioning Score at Treatment Discontinuation Visit: number analyzed (Participants) | 114 | 46
  Emotional functioning Score at Treatment Discontinuation Visit | 63.6 (28.2) | 70.3 (23.2)
  Emotional functioning Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Emotional functioning Score at 30-Day Safety Follow-up | 70.5 (24.7) | 82.0 (17.4)
  Social functioning Score at Screening: number analyzed (Participants) | 223 | 111
  Social functioning Score at Screening | 79.9 (23.9) | 79.0 (24.8)
  Social functioning Score at Week 9: number analyzed (Participants) | 179 | 82
  Social functioning Score at Week 9 | 69.5 (26.0) | 76.2 (28.0)
  Social functioning Score at Week 17: number analyzed (Participants) | 136 | 68
  Social functioning Score at Week 17 | 75.6 (21.8) | 77.7 (23.9)
  Social functioning Score at Week 25: number analyzed (Participants) | 109 | 47
  Social functioning Score at Week 25 | 78.7 (21.3) | 76.6 (23.2)
  Social functioning Score at Week 33: number analyzed (Participants) | 86 | 31
  Social functioning Score at Week 33 | 76.0 (23.8) | 79.0 (26.5)
  Social functioning Score at Week 41: number analyzed (Participants) | 77 | 25
  Social functioning Score at Week 41 | 73.4 (25.0) | 83.3 (25.5)
  Social functioning Score at Week 49: number analyzed (Participants) | 65 | 18
  Social functioning Score at Week 49 | 78.5 (20.6) | 81.5 (16.1)
  Social functioning Score at Week 57: number analyzed (Participants) | 43 | 16
  Social functioning Score at Week 57 | 74.0 (24.2) | 77.1 (27.1)
  Social functioning Score at Week 65: number analyzed (Participants) | 40 | 11
  Social functioning Score at Week 65 | 78.3 (23.9) | 72.7 (31.9)
  Social functioning Score at Week 73: number analyzed (Participants) | 34 | 8
  Social functioning Score at Week 73 | 75.5 (25.4) | 75.0 (28.2)
  Social functioning Score at Treatment Discontinuation Visit: number analyzed (Participants) | 114 | 46
  Social functioning Score at Treatment Discontinuation Visit | 63.5 (32.7) | 66.7 (31.2)
  Social functioning Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Social functioning Score at 30-Day Safety Follow-up | 71.1 (27.9) | 78.1 (27.2)

9. Secondary Outcome: Quality of Life Per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Ovarian Cancer Module (QLQ-OV28)
Description: EORTC QLQ-OV28 contains 28 items which assess a comprehensive range of relevant issues: abdominal/gastrointestinal (GI) symptoms, peripheral neuropathy, other chemotherapy side-effects, hormonal/menopausal symptoms, body image, attitude to disease/treatment and sexual functioning. The score for each domain and component score were scaled from 0 (minimum) to 100 (maximum). Higher scores indicate lower quality of life except for sexual functioning where higher scores indicate better quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MEK 162 | Physician's Choice
Number analyzed (Participants) | 228 | 113
Scores on a scale
  Abdominal/GI Score at Screening: number analyzed (Participants) | 220 | 111
  Abdominal/GI Score at Screening | 22.8 (18.6) | 25.7 (22.5)
  Abdominal/GI Score at Week 9: number analyzed (Participants) | 171 | 81
  Abdominal/GI Score at Week 9 | 29.3 (20.1) | 22.3 (17.7)
  Abdominal/GI Score at Week 17: number analyzed (Participants) | 134 | 67
  Abdominal/GI Score at Week 17 | 26.7 (19.6) | 20.3 (15.9)
  Abdominal/GI Score at Week 25: number analyzed (Participants) | 108 | 46
  Abdominal/GI Score at Week 25 | 22.1 (18.6) | 20.9 (17.2)
  Abdominal/GI Score at Week 33: number analyzed (Participants) | 86 | 32
  Abdominal/GI Score at Week 33 | 27.2 (20.3) | 15.6 (18.3)
  Abdominal/GI Score at Week 41: number analyzed (Participants) | 76 | 25
  Abdominal/GI Score at Week 41 | 26.9 (20.3) | 18.7 (23.0)
  Abdominal/GI Score at Week 49: number analyzed (Participants) | 64 | 18
  Abdominal/GI Score at Week 49 | 23.5 (20.5) | 17.6 (20.7)
  Abdominal/GI Score at Week 57: number analyzed (Participants) | 43 | 16
  Abdominal/GI Score at Week 57 | 26.1 (20.4) | 18.4 (19.3)
  Abdominal/GI Score at Week 65: number analyzed (Participants) | 41 | 11
  Abdominal/GI Score at Week 65 | 26.0 (19.4) | 23.7 (23.1)
  Abdominal/GI Score at Week 73: number analyzed (Participants) | 33 | 8
  Abdominal/GI Score at Week 73 | 23.0 (20.3) | 31.3 (29.1)
  Abdominal/GI Score at Treatment Discontinuation Visit: number analyzed (Participants) | 109 | 45
  Abdominal/GI Score at Treatment Discontinuation Visit | 31.6 (22.0) | 24.1 (20.4)
  Abdominal/GI Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Abdominal/GI Score at 30-Day Safety Follow-up | 31.8 (24.6) | 17.5 (22.1)
  Peripheral neuropathy Score at Screening: number analyzed (Participants) | 220 | 110
  Peripheral neuropathy Score at Screening | 16.6 (26.1) | 14.5 (22.4)
  Peripheral neuropathy Score at Week 9: number analyzed (Participants) | 171 | 81
  Peripheral neuropathy Score at Week 9 | 26.7 (29.9) | 19.5 (23.5)
  Peripheral neuropathy Score at Week 17: number analyzed (Participants) | 134 | 67
  Peripheral neuropathy Score at Week 17 | 27.1 (28.8) | 20.9 (21.6)
  Peripheral neuropathy Score at Week 25: number analyzed (Participants) | 108 | 46
  Peripheral neuropathy Score at Week 25 | 30.2 (31.0) | 21.0 (24.2)
  Peripheral neuropathy Score at Week 33: number analyzed (Participants) | 86 | 32
  Peripheral neuropathy Score at Week 33 | 30.4 (28.7) | 21.4 (24.4)
  Peripheral neuropathy Score at Week 41: number analyzed (Participants) | 76 | 25
  Peripheral neuropathy Score at Week 41 | 25.2 (30.1) | 14.0 (16.4)
  Peripheral neuropathy Score at Week 49: number analyzed (Participants) | 64 | 18
  Peripheral neuropathy Score at Week 49 | 25.0 (24.1) | 16.7 (18.1)
  Peripheral neuropathy Score at Week 57: number analyzed (Participants) | 43 | 16
  Peripheral neuropathy Score at Week 57 | 22.5 (27.9) | 15.6 (23.9)
  Peripheral neuropathy Score at Week 65: number analyzed (Participants) | 41 | 11
  Peripheral neuropathy Score at Week 65 | 18.7 (24.8) | 22.7 (26.1)
  Peripheral neuropathy Score at Week 73: number analyzed (Participants) | 33 | 8
  Peripheral neuropathy Score at Week 73 | 17.2 (27.2) | 25.0 (30.9)
  Peripheral neuropathy Score at Treatment Discontinuation Visit: number analyzed (Participants) | 108 | 45
  Peripheral neuropathy Score at Treatment Discontinuation Visit | 28.5 (32.4) | 22.6 (24.4)
  Peripheral neuropathy Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Peripheral neuropathy Score at 30-Day Safety Follow-up | 28.9 (29.8) | 23.7 (32.5)
  Hormonal Score at Screening: number analyzed (Participants) | 220 | 110
  Hormonal Score at Screening | 22.0 (25.5) | 23.3 (28.4)
  Hormonal Score at Week 9: number analyzed (Participants) | 171 | 81
  Hormonal Score at Week 9 | 10.2 (15.5) | 23.7 (28.9)
  Hormonal Score at Week 17: number analyzed (Participants) | 134 | 67
  Hormonal Score at Week 17 | 9.3 (16.8) | 23.1 (28.1)
  Hormonal Score at Week 25: number analyzed (Participants) | 108 | 46
  Hormonal Score at Week 25 | 6.2 (11.5) | 23.2 (26.2)
  Hormonal Score at Week 33: number analyzed (Participants) | 86 | 32
  Hormonal Score at Week 33 | 11.6 (20.0) | 23.4 (29.0)
  Hormonal Score at Week 41: number analyzed (Participants) | 76 | 25
  Hormonal Score at Week 41 | 13.4 (22.9) | 21.3 (29.9)
  Hormonal Score at Week 49: number analyzed (Participants) | 64 | 18
  Hormonal Score at Week 49 | 13.8 (22.3) | 25.9 (34.4)
  Hormonal Score at Week 57: number analyzed (Participants) | 43 | 16
  Hormonal Score at Week 57 | 11.2 (16.6) | 33.3 (38.0)
  Hormonal Score at Week 65: number analyzed (Participants) | 41 | 11
  Hormonal Score at Week 65 | 9.8 (15.8) | 25.8 (38.3)
  Hormonal Score at Week 73: number analyzed (Participants) | 33 | 8
  Hormonal Score at Week 73 | 8.1 (13.3) | 14.6 (28.8)
  Hormonal Score at Treatment Discontinuation Visit: number analyzed (Participants) | 108 | 45
  Hormonal Score at Treatment Discontinuation Visit | 14.8 (21.7) | 26.7 (34.0)
  Hormonal Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Hormonal Score at 30-Day Safety Follow-up | 22.4 (27.8) | 14.9 (21.4)
  Body image Score at Screening: number analyzed (Participants) | 217 | 111
  Body image Score at Screening | 28.9 (29.3) | 31.4 (31.9)
  Body image Score at Week 9: number analyzed (Participants) | 170 | 80
  Body image Score at Week 9 | 42.1 (32.1) | 36.0 (30.1)
  Body image Score at Week 17: number analyzed (Participants) | 133 | 67
  Body image Score at Week 17 | 40.1 (29.6) | 32.6 (29.9)
  Body image Score at Week 25: number analyzed (Participants) | 107 | 47
  Body image Score at Week 25 | 37.4 (29.1) | 27.7 (25.4)
  Body image Score at Week 33: number analyzed (Participants) | 86 | 32
  Body image Score at Week 33 | 36.2 (25.7) | 28.6 (29.1)
  Body image Score at Week 41: number analyzed (Participants) | 76 | 25
  Body image Score at Week 41 | 40.4 (26.8) | 30.0 (31.2)
  Body image Score at Week 49: number analyzed (Participants) | 64 | 18
  Body image Score at Week 49 | 36.2 (25.8) | 25.9 (32.5)
  Body image Score at Week 57: number analyzed (Participants) | 42 | 16
  Body image Score at Week 57 | 36.1 (27.0) | 16.7 (26.5)
  Body image Score at Week 65: number analyzed (Participants) | 41 | 11
  Body image Score at Week 65 | 33.7 (28.0) | 25.8 (30.2)
  Body image Score at Week 73: number analyzed (Participants) | 33 | 8
  Body image Score at Week 73 | 27.8 (23.4) | 33.3 (34.5)
  Body image Score at Treatment Discontinuation Visit: number analyzed (Participants) | 109 | 45
  Body image Score at Treatment Discontinuation Visit | 46.9 (32.9) | 37.0 (32.0)
  Body image Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Body image Score at 30-Day Safety Follow-up | 35.0 (30.5) | 23.7 (26.8)
  Attitude to disease/treatment Score at Screening: number analyzed (Participants) | 216 | 110
  Attitude to disease/treatment Score at Screening | 48.0 (28.6) | 51.4 (29.1)
  Attitude to disease/treatment Score at Week 9: number analyzed (Participants) | 169 | 80
  Attitude to disease/treatment Score at Week 9 | 49.5 (25.5) | 47.6 (26.5)
  Attitude to disease/treatment Score at Week 17: number analyzed (Participants) | 133 | 67
  Attitude to disease/treatment Score at Week 17 | 46.1 (24.2) | 51.6 (26.1)
  Attitude to disease/treatment Score at Week 25: number analyzed (Participants) | 107 | 47
  Attitude to disease/treatment Score at Week 25 | 39.0 (22.2) | 44.1 (26.5)
  Attitude to disease/treatment Score at Week 33: number analyzed (Participants) | 86 | 32
  Attitude to disease/treatment Score at Week 33 | 41.8 (22.9) | 44.4 (24.8)
  Attitude to disease/treatment Score at Week 41: number analyzed (Participants) | 76 | 25
  Attitude to disease/treatment Score at Week 41 | 44.3 (23.1) | 40.4 (23.1)
  Attitude to disease/treatment Score at Week 49: number analyzed (Participants) | 64 | 18
  Attitude to disease/treatment Score at Week 49 | 37.2 (19.7) | 38.9 (23.6)
  Attitude to disease/treatment Score at Week 57: number analyzed (Participants) | 42 | 16
  Attitude to disease/treatment Score at Week 57 | 38.8 (20.0) | 32.6 (27.1)
  Attitude to disease/treatment Score at Week 65: number analyzed (Participants) | 41 | 11
  Attitude to disease/treatment Score at Week 65 | 37.4 (21.6) | 45.5 (28.7)
  Attitude to disease/treatment Score at Week 73: number analyzed (Participants) | 33 | 8
  Attitude to disease/treatment Score at Week 73 | 37.7 (25.3) | 51.4 (43.6)
  Attitude to disease/treatment Score at Treatment Discontinuation Visit: number analyzed (Participants) | 109 | 45
  Attitude to disease/treatment Score at Treatment Discontinuation Visit | 55.8 (27.5) | 53.8 (29.3)
  Attitude to disease/treatment Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Attitude to disease/treatment Score at 30-Day Safety Follow-up | 49.3 (27.0) | 50.3 (24.9)
  Chemotherapy Side Effects Score at Screening: number analyzed (Participants) | 220 | 110
  Chemotherapy Side Effects Score at Screening | 17.7 (16.0) | 17.1 (14.7)
  Chemotherapy Side Effects Score at Week 9: number analyzed (Participants) | 171 | 81
  Chemotherapy Side Effects Score at Week 9 | 28.6 (16.4) | 22.6 (16.2)
  Chemotherapy Side Effects Score at Week 17: number analyzed (Participants) | 134 | 67
  Chemotherapy Side Effects Score at Week 17 | 27.1 (15.3) | 24.1 (15.2)
  Chemotherapy Side Effects Score at Week 25: number analyzed (Participants) | 108 | 46
  Chemotherapy Side Effects Score at Week 25 | 27.7 (17.5) | 25.3 (18.1)
  Chemotherapy Side Effects Score at Week 33: number analyzed (Participants) | 86 | 32
  Chemotherapy Side Effects Score at Week 33 | 28.8 (18.4) | 24.1 (17.1)
  Chemotherapy Side Effects Score at Week 41: number analyzed (Participants) | 75 | 25
  Chemotherapy Side Effects Score at Week 41 | 30.1 (19.2) | 23.5 (20.8)
  Chemotherapy Side Effects Score at Week 49: number analyzed (Participants) | 64 | 18
  Chemotherapy Side Effects Score at Week 49 | 29.5 (16.5) | 23.0 (18.6)
  Chemotherapy Side Effects Score at Week 57: number analyzed (Participants) | 43 | 16
  Chemotherapy Side Effects Score at Week 57 | 27.9 (19.5) | 23.1 (18.3)
  Chemotherapy Side Effects Score at Week 65: number analyzed (Participants) | 41 | 11
  Chemotherapy Side Effects Score at Week 65 | 25.5 (19.1) | 25.5 (15.4)
  Chemotherapy Side Effects Score at Week 73: number analyzed (Participants) | 33 | 8
  Chemotherapy Side Effects Score at Week 73 | 27.7 (19.4) | 29.2 (20.5)
  Chemotherapy Side Effects Score at Treatment Discontinuation Visit: number analyzed (Participants) | 108 | 45
  Chemotherapy Side Effects Score at Treatment Discontinuation Visit | 30.4 (19.6) | 28.0 (19.4)
  Chemotherapy Side Effects Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Chemotherapy Side Effects Score at 30-Day Safety Follow-up | 27.5 (19.5) | 17.9 (14.7)
  Other Score at Screening: number analyzed (Participants) | 220 | 111
  Other Score at Screening | 11.8 (16.5) | 14.5 (19.6)
  Other Score at Week 9: number analyzed (Participants) | 171 | 81
  Other Score at Week 9 | 22.0 (17.4) | 23.3 (20.6)
  Other Score at Week 17: number analyzed (Participants) | 134 | 67
  Other Score at Week 17 | 26.1 (22.2) | 20.1 (19.1)
  Other Score at Week 25: number analyzed (Participants) | 108 | 46
  Other Score at Week 25 | 22.9 (21.1) | 18.7 (17.5)
  Other Score at Week 33: number analyzed (Participants) | 86 | 32
  Other Score at Week 33 | 22.3 (21.3) | 16.7 (19.4)
  Other Score at Week 41: number analyzed (Participants) | 76 | 25
  Other Score at Week 41 | 19.1 (20.2) | 14.3 (15.1)
  Other Score at Week 49: number analyzed (Participants) | 64 | 18
  Other Score at Week 49 | 19.0 (18.6) | 12.8 (13.6)
  Other Score at Week 57: number analyzed (Participants) | 43 | 16
  Other Score at Week 57 | 16.3 (15.5) | 16.8 (17.0)
  Other Score at Week 65: number analyzed (Participants) | 41 | 11
  Other Score at Week 65 | 15.4 (12.9) | 22.0 (24.5)
  Other Score at Week 73: number analyzed (Participants) | 33 | 8
  Other Score at Week 73 | 15.7 (15.0) | 22.2 (22.0)
  Other Score at Treatment Discontinuation Visit: number analyzed (Participants) | 109 | 45
  Other Score at Treatment Discontinuation Visit | 22.1 (16.9) | 22.7 (20.1)
  Other Score at 30-Day Safety Follow-up: number analyzed (Participants) | 41 | 19
  Other Score at 30-Day Safety Follow-up | 17.2 (17.0) | 14.6 (20.4)
  Sexuality Score at Screening: number analyzed (Participants) | 200 | 106
  Sexuality Score at Screening | 20.2 (20.3) | 19.2 (21.9)
  Sexuality Score at Week 9: number analyzed (Participants) | 151 | 78
  Sexuality Score at Week 9 | 18.7 (20.4) | 18.1 (21.9)
  Sexuality Score at Week 17: number analyzed (Participants) | 113 | 65
  Sexuality Score at Week 17 | 19.6 (20.3) | 18.3 (21.6)
  Sexuality Score at Week 25: number analyzed (Participants) | 91 | 44
  Sexuality Score at Week 25 | 21.8 (21.5) | 22.0 (23.8)
  Sexuality Score at Week 33: number analyzed (Participants) | 75 | 29
  Sexuality Score at Week 33 | 25.8 (23.0) | 21.3 (21.7)
  Sexuality Score at Week 41: number analyzed (Participants) | 68 | 23
  Sexuality Score at Week 41 | 21.3 (20.0) | 19.2 (23.1)
  Sexuality Score at Week 49: number analyzed (Participants) | 57 | 17
  Sexuality Score at Week 49 | 23.0 (21.9) | 20.6 (23.0)
  Sexuality Score at Week 57: number analyzed (Participants) | 37 | 15
  Sexuality Score at Week 57 | 21.8 (21.8) | 18.9 (24.7)
  Sexuality Score at Week 65: number analyzed (Participants) | 36 | 10
  Sexuality Score at Week 65 | 21.3 (20.7) | 12.5 (15.8)
  Sexuality Score at Week 73: number analyzed (Participants) | 30 | 7
  Sexuality Score at Week 73 | 20.8 (21.6) | 11.9 (16.6)
  Sexuality Score at Treatment Discontinuation Visit: number analyzed (Participants) | 95 | 42
  Sexuality Score at Treatment Discontinuation Visit | 14.2 (19.4) | 23.2 (23.0)
  Sexuality Score at 30-Day Safety Follow-up: number analyzed (Participants) | 38 | 18
  Sexuality Score at 30-Day Safety Follow-up | 15.6 (19.8) | 26.1 (25.8)

10. Secondary Outcome: Quality of Life Per Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-NTX)
Description: FACT/GOG-NTX questionnaire consists of questions for dimensions related to physical, social, emotional, and functional well-being which contains 11 items, with responses scored on a Likert scale from 0 (not at all) to 4 (very much) designed to capture the symptoms of chemotherapy-induced peripheral neuropathy (CIPN). The summed scores of each item were reverted into standardized scores ranging from 0 to 44, with a higher score indicating a lower level of neurological toxicity and less effect on quality of life (ie, higher scores indicate better quality of life). The trial outcome index consists of two subscales from the FACT-G: Physical Well Being (7 items) and Functional Well Being (7 items), plus the Cervix Cancer-specific subscale (15 items). Each item in the trial outcome index scored using a 5-point scale (0=not at all to 4=very much). The summed scores of each item were reverted into standardized scores ranging from 0 to 116. Higher scores indicate better quality of life.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MEK 162 | Physician's Choice
Number analyzed (Participants) | 228 | 113
Scores on a scale
  Physical Well-being Score at Screening: number analyzed (Participants) | 218 | 111
  Physical Well-being Score at Screening | 21.7 (5.1) | 21.6 (5.7)
  Physical Well-being Score at Week 9: number analyzed (Participants) | 173 | 81
  Physical Well-being Score at Week 9 | 19.0 (5.7) | 21.4 (5.5)
  Physical Well-being Score at Week 17: number analyzed (Participants) | 134 | 67
  Physical Well-being Score at Week 17 | 20.1 (4.9) | 21.5 (5.2)
  Physical Well-being Score at Week 25: number analyzed (Participants) | 106 | 46
  Physical Well-being Score at Week 25 | 20.4 (5.2) | 21.3 (6.1)
  Physical Well-being Score at Week 33: number analyzed (Participants) | 85 | 32
  Physical Well-being Score at Week 33 | 20.2 (5.1) | 21.2 (6.3)
  Physical Well-being Score at Week 41: number analyzed (Participants) | 76 | 25
  Physical Well-being Score at Week 41 | 19.9 (5.5) | 22.6 (6.6)
  Physical Well-being Score at Week 49: number analyzed (Participants) | 63 | 18
  Physical Well-being Score at Week 49 | 20.5 (4.9) | 22.6 (6.2)
  Physical Well-being Score at Week 57: number analyzed (Participants) | 42 | 16
  Physical Well-being Score at Week 57 | 20.8 (4.6) | 22.4 (6.1)
  Physical Well-being Score at Week 65: number analyzed (Participants) | 39 | 11
  Physical Well-being Score at Week 65 | 21.3 (4.7) | 20.2 (7.2)
  Physical Well-being Score at Week 73: number analyzed (Participants) | 31 | 8
  Physical Well-being Score at Week 73 | 21.8 (4.5) | 20.8 (8.4)
  Physical Well-being Score at Treatment Discontinuation Visit: number analyzed (Participants) | 107 | 46
  Physical Well-being Score at Treatment Discontinuation Visit | 17.8 (6.7) | 19.4 (7.4)
  Physical Well-being Score at 30-Day Safety Follow-up: number analyzed (Participants) | 40 | 18
  Physical Well-being Score at 30-Day Safety Follow-up | 19.6 (6.5) | 23.1 (4.7)
  Social Well-being Score at Screening: number analyzed (Participants) | 216 | 111
  Social Well-being Score at Screening | 20.7 (4.8) | 20.7 (4.9)
  Social Well-being Score at Week 9: number analyzed (Participants) | 172 | 81
  Social Well-being Score at Week 9 | 20.0 (4.6) | 20.3 (5.0)
  Social Well-being Score at Week 17: number analyzed (Participants) | 134 | 67
  Social Well-being Score at Week 17 | 19.7 (5.1) | 20.6 (4.4)
  Social Well-being Score at Week 25: number analyzed (Participants) | 105 | 46
  Social Well-being Score at Week 25 | 20.3 (4.6) | 20.2 (4.6)
  Social Well-being Score at Week 33: number analyzed (Participants) | 85 | 32
  Social Well-being Score at Week 33 | 20.3 (5.5) | 21.0 (5.0)
  Social Well-being Score at Week 41: number analyzed (Participants) | 76 | 25
  Social Well-being Score at Week 41 | 20.7 (5.0) | 21.3 (4.9)
  Social Well-being Score at Week 49: number analyzed (Participants) | 63 | 18
  Social Well-being Score at Week 49 | 20.6 (4.6) | 21.4 (4.8)
  Social Well-being Score at Week 57: number analyzed (Participants) | 42 | 16
  Social Well-being Score at Week 57 | 20.0 (5.9) | 21.5 (5.1)
  Social Well-being Score at Week 65: number analyzed (Participants) | 39 | 11
  Social Well-being Score at Week 65 | 20.5 (5.4) | 20.6 (5.4)
  Social Well-being Score at Week 73: number analyzed (Participants) | 31 | 8
  Social Well-being Score at Week 73 | 20.0 (6.1) | 22.1 (5.0)
  Peripheral neuropathy Score at Treatment Discontinuation Visit: number analyzed (Participants) | 107 | 46
  Peripheral neuropathy Score at Treatment Discontinuation Visit | 19.3 (4.7) | 20.7 (4.5)
  Peripheral neuropathy Score at 30-Day Safety Follow-up: number analyzed (Participants) | 40 | 18
  Peripheral neuropathy Score at 30-Day Safety Follow-up | 20.5 (4.3) | 21.0 (4.9)
  Emotional Well-being Score at Screening: number analyzed (Participants) | 217 | 110
  Emotional Well-being Score at Screening | 16.1 (5.1) | 15.4 (5.0)
  Emotional Well-being Score at Week 9: number analyzed (Participants) | 171 | 81
  Emotional Well-being Score at Week 9 | 16.5 (4.7) | 16.4 (4.7)
  Emotional Well-being Score at Week 17: number analyzed (Participants) | 132 | 67
  Emotional Well-being Score at Week 17 | 17.2 (4.2) | 17.0 (4.1)
  Emotional Well-being Score at Week 25: number analyzed (Participants) | 104 | 46
  Emotional Well-being Score at Week 25 | 17.3 (4.4) | 17.5 (3.9)
  Emotional Well-being Score at Week 33: number analyzed (Participants) | 85 | 32
  Emotional Well-being Score at Week 33 | 17.3 (4.3) | 18.0 (4.8)
  Emotional Well-being Score at Week 41: number analyzed (Participants) | 75 | 25
  Emotional Well-being Score at Week 41 | 16.9 (4.4) | 18.0 (4.9)
  Emotional Well-being Score at Week 49: number analyzed (Participants) | 64 | 18
  Emotional Well-being Score at Week 49 | 17.4 (3.8) | 18.1 (4.6)
  Emotional Well-being Score at Week 57: number analyzed (Participants) | 43 | 16
  Emotional Well-being Score at Week 57 | 17.5 (4.1) | 19.2 (3.2)
  Emotional Well-being Score at Week 65: number analyzed (Participants) | 40 | 11
  Emotional Well-being Score at Week 65 | 18.1 (3.8) | 17.7 (3.6)
  Emotional Well-being Score at Week 73: number analyzed (Participants) | 30 | 8
  Emotional Well-being Score at Week 73 | 18.3 (3.2) | 17.3 (5.8)
  Emotional Well-being Score at Treatment Discontinuation Visit: number analyzed (Participants) | 106 | 46
  Emotional Well-being Score at Treatment Discontinuation Visit | 14.5 (5.9) | 15.4 (5.6)
  Emotional Well-being Score at 30-Day Safety Follow-up: number analyzed (Participants) | 39 | 18
  Emotional Well-being Score at 30-Day Safety Follow-up | 15.4 (5.4) | 17.3 (4.7)
  Functional Well-being Score at Screening: number analyzed (Participants) | 217 | 111
  Functional Well-being Score at Screening | 18.0 (6.0) | 18.3 (6.5)
  Functional Well-being Score at Week 9: number analyzed (Participants) | 172 | 81
  Functional Well-being Score at Week 9 | 16.2 (6.2) | 18.1 (6.0)
  Functional Well-being Score at Week 17: number analyzed (Participants) | 132 | 67
  Functional Well-being Score at Week 17 | 16.9 (5.7) | 17.3 (5.8)
  Functional Well-being Score at Week 25: number analyzed (Participants) | 105 | 46
  Functional Well-being Score at Week 25 | 17.4 (5.3) | 17.7 (5.8)
  Functional Well-being Score at Week 33: number analyzed (Participants) | 85 | 32
  Functional Well-being Score at Week 33 | 17.5 (5.7) | 18.8 (6.1)
  Functional Well-being Score at Week 41: number analyzed (Participants) | 75 | 25
  Functional Well-being Score at Week 41 | 17.5 (5.3) | 19.8 (7.4)
  Functional Well-being Score at Week 49: number analyzed (Participants) | 64 | 18
  Functional Well-being Score at Week 49 | 18.0 (5.0) | 19.1 (6.3)
  Functional Well-being Score at Week 57: number analyzed (Participants) | 43 | 16
  Functional Well-being Score at Week 57 | 17.0 (6.3) | 20.4 (6.6)
  Functional Well-being Score at Week 65: number analyzed (Participants) | 40 | 11
  Functional Well-being Score at Week 65 | 18.3 (5.7) | 18.9 (6.1)
  Functional Well-being Score at Week 73: number analyzed (Participants) | 30 | 8
  Functional Well-being Score at Week 73 | 18.7 (5.4) | 19.8 (5.8)
  Functional Well-being Score at Treatment Discontinuation Visit: number analyzed (Participants) | 106 | 46
  Functional Well-being Score at Treatment Discontinuation Visit | 15.0 (6.0) | 17.0 (7.0)
  Functional Well-being Score at 30-Day Safety Follow-up: number analyzed (Participants) | 39 | 18
  Functional Well-being Score at 30-Day Safety Follow-up | 16.5 (6.1) | 18.8 (6.5)
  Neurotoxicity Subscale Score at Screening: number analyzed (Participants) | 217 | 111
  Neurotoxicity Subscale Score at Screening | 38.0 (6.4) | 39.0 (6.0)
  Neurotoxicity Subscale Score at Week 9: number analyzed (Participants) | 172 | 81
  Neurotoxicity Subscale Score at Week 9 | 36.2 (6.5) | 37.8 (6.4)
  Neurotoxicity Subscale Score at Week 17: number analyzed (Participants) | 131 | 67
  Neurotoxicity Subscale Score at Week 17 | 35.9 (7.1) | 37.1 (5.9)
  Neurotoxicity Subscale Score at Week 25: number analyzed (Participants) | 105 | 46
  Neurotoxicity Subscale Score at Week 25 | 35.1 (7.6) | 36.6 (6.1)
  Neurotoxicity Subscale Score at Week 33: number analyzed (Participants) | 85 | 32
  Neurotoxicity Subscale Score at Week 33 | 35.2 (6.8) | 36.6 (7.5)
  Neurotoxicity Subscale Score at Week 41: number analyzed (Participants) | 74 | 25
  Neurotoxicity Subscale Score at Week 41 | 35.6 (7.2) | 37.7 (5.9)
  Neurotoxicity Subscale Score at Week 49: number analyzed (Participants) | 65 | 18
  Neurotoxicity Subscale Score at Week 49 | 35.1 (7.1) | 37.6 (7.9)
  Neurotoxicity Subscale Score at Week 57: number analyzed (Participants) | 43 | 16
  Neurotoxicity Subscale Score at Week 57 | 35.9 (7.3) | 37.3 (7.4)
  Neurotoxicity Subscale Score at Week 65: number analyzed (Participants) | 40 | 11
  Neurotoxicity Subscale Score at Week 65 | 36.6 (7.4) | 35.5 (7.1)
  Neurotoxicity Subscale Score at Week 73: number analyzed (Participants) | 30 | 8
  Neurotoxicity Subscale Score at Week 73 | 37.5 (6.7) | 34.3 (8.8)
  Neurotoxicity Subscale Score at Treatment Discontinuation Visit: number analyzed (Participants) | 106 | 45
  Neurotoxicity Subscale Score at Treatment Discontinuation Visit | 34.6 (7.8) | 36.0 (7.3)
  Neurotoxicity Subscale Score at 30-Day Safety Follow-up: number analyzed (Participants) | 39 | 18
  Neurotoxicity Subscale Score at 30-Day Safety Follow-up | 34.7 (9.0) | 37.8 (7.5)
  Trial Outcome Index Score at Screening: number analyzed (Participants) | 215 | 111
  Trial Outcome Index Score at Screening | 78.0 (13.6) | 78.9 (15.3)
  Trial Outcome Index Score at Week 9: number analyzed (Participants) | 169 | 81
  Trial Outcome Index Score at Week 9 | 71.5 (14.4) | 77.3 (15.2)
  Trial Outcome Index Score at Week 17: number analyzed (Participants) | 131 | 67
  Trial Outcome Index Score at Week 17 | 72.9 (13.5) | 76.0 (14.2)
  Trial Outcome Index Score at Week 25: number analyzed (Participants) | 105 | 46
  Trial Outcome Index Score at Week 25 | 72.8 (15.0) | 75.7 (16.1)
  Trial Outcome Index Score at Week 33: number analyzed (Participants) | 85 | 32
  Trial Outcome Index Score at Week 33 | 72.9 (14.7) | 76.6 (17.4)
  Trial Outcome Index Score at Week 41: number analyzed (Participants) | 74 | 25
  Trial Outcome Index Score at Week 41 | 73.3 (13.8) | 80.1 (18.0)
  Trial Outcome Index Score at Week 49: number analyzed (Participants) | 63 | 18
  Trial Outcome Index Score at Week 49 | 74.1 (13.4) | 79.3 (17.6)
  Trial Outcome Index Score at Week 57: number analyzed (Participants) | 42 | 16
  Trial Outcome Index Score at Week 57 | 74.4 (13.9) | 80.1 (17.1)
  Trial Outcome Index Score at Week 65: number analyzed (Participants) | 39 | 11
  Trial Outcome Index Score at Week 65 | 77.2 (13.5) | 74.6 (16.4)
  Trial Outcome Index Score at Week 73: number analyzed (Participants) | 30 | 8
  Trial Outcome Index Score at Week 73 | 77.9 (14.2) | 74.8 (20.9)
  Trial Outcome Index Score at Treatment Discontinuation Visit: number analyzed (Participants) | 106 | 45
  Trial Outcome Index Score at Treatment Discontinuation Visit | 67.5 (16.5) | 72.1 (18.0)
  Trial Outcome Index Score at 30-Day Safety Follow-up: number analyzed (Participants) | 39 | 18
  Trial Outcome Index Score at 30-Day Safety Follow-up | 70.8 (17.5) | 79.8 (15.7)

11. Secondary Outcome: Predose Plasma Concentration (Ctrough) of MEK162
Description: Ctrough of MEK162 is defined as the predose plasma concentration of MEK162. Ctrough of MEK162 was observed directly from data.
Time Frame: Predose on Study Days 1, 57, and 113.
Population: The pharmacokinetics (PK) set consisted of all participants who received at least 1 dose of MEK162 and had at least 1 PK blood collection with associated bioanalytical results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | MEK162
Number analyzed (Participants) | 65
nanograms per milliliter (ng/mL)
  Week 1 (Study Day 1) | 42.2 (NA) — The geometric coefficient of variation was statistically non-estimable for this dataset at Week 1 (Study Day 1).
  Week 9 (Study Day 57): number analyzed (Participants) | 38
  Week 9 (Study Day 57) | 69.3 (1.54)
  Week 17 (Study Day 113): number analyzed (Participants) | 33
  Week 17 (Study Day 113) | 56.5 (1.68)

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MEK162
Description: Cmax is maximum observed plasma concentration. Cmax of MEK162 was observed directly from data.
Time Frame: 2 hours ± 10 minutes postdose on Study Days 1, 57, and 113.
Population: The PK set consisted of all participants who received at least 1 dose of MEK162 and had at least 1 PK blood collection with associated bioanalytical results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MEK162
Number analyzed (Participants) | 52
ng/mL
  Week 1 (Study Day 1) | 339 (0.544)
  Week 9 (Study Day 57): number analyzed (Participants) | 30
  Week 9 (Study Day 57) | 343 (0.959)
  Week 17 (Study Day 113): number analyzed (Participants) | 20
  Week 17 (Study Day 113) | 304 (0.649)

ADVERSE EVENTS:
Time Frame: From the first dose of study intervention until 30 days after the last dose (up to 9 years)
Description: Same event might appear as AE and serious AE, what was presented are distinct events. Event might be categorized as serious in 1 participant and as non-serious in another or 1 participant might have experienced both during study. Safety set included all participants who received at least 1 dose of study intervention and have at least 1 post-treatment assessment, including death. Crossover set all-cause mortality and AEs were not collected given the early stopping of the crossover period.
Arm/Group | MEK162 | Physician's Choice
All-Cause Mortality (participants affected / at risk) | 89/227 | 42/106
Serious Adverse Events (participants affected / at risk) | 126/227 | 31/106
Other Adverse Events (participants affected / at risk) | 226/227 | 105/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MEK162 (N=227) | Physician's Choice (N=106)
Small intestinal obstruction (Gastrointestinal disorders) | 12 | 8
Vomiting (Gastrointestinal disorders) | 16 | 2
Intestinal obstruction (Gastrointestinal disorders) | 15 | 4
Ascites (Gastrointestinal disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 10 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 2
Nausea (Gastrointestinal disorders) | 7 | 1
Colonic obstruction (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Subileus (Gastrointestinal disorders) | 7 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 9 | 1
Urinary tract infection (Infections and infestations) | 8 | 1
Lung infection (Infections and infestations) | 3 | 0
Device related infection (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 4 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection fungal (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death (General disorders) | 3 | 1
Asthenia (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 9 | 2
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 4 | 0
Ejection fraction decreased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 2 | 0
Troponin I increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Retinal vein occlusion (Eye disorders) | 4 | 0
Choroiditis (Eye disorders) | 1 | 0
Retinal oedema (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 6 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dropped head syndrome (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Panic reaction (Psychiatric disorders) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Ileal fistula (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 1
Generalised oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Psoas abscess (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 2 | 0
Aspiration pleural cavity (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MEK162 (N=227) | Physician's Choice (N=106)
Diarrhoea (Gastrointestinal disorders) | 160 | 39
Nausea (Gastrointestinal disorders) | 135 | 55
Vomiting (Gastrointestinal disorders) | 129 | 32
Abdominal pain (Gastrointestinal disorders) | 77 | 27
Constipation (Gastrointestinal disorders) | 66 | 31
Stomatitis (Gastrointestinal disorders) | 54 | 35
Dyspepsia (Gastrointestinal disorders) | 32 | 11
Dry mouth (Gastrointestinal disorders) | 37 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 | 7
Abdominal distension (Gastrointestinal disorders) | 25 | 6
Abdominal pain upper (Gastrointestinal disorders) | 23 | 6
Ascites (Gastrointestinal disorders) | 15 | 6
Rectal haemorrhage (Gastrointestinal disorders) | 10 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 110 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 57 | 28
Dry skin (Skin and subcutaneous tissue disorders) | 77 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 57 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 51 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 | 36
Rash (Skin and subcutaneous tissue disorders) | 36 | 10
Skin fissures (Skin and subcutaneous tissue disorders) | 34 | 1
Fatigue (General disorders) | 120 | 54
Oedema peripheral (General disorders) | 120 | 16
Pyrexia (General disorders) | 42 | 17
Asthenia (General disorders) | 29 | 7
Face oedema (General disorders) | 28 | 1
Chills (General disorders) | 16 | 5
Non-cardiac chest pain (General disorders) | 11 | 7
Blood creatine phosphokinase increased (Investigations) | 120 | 2
Ejection fraction decreased (Investigations) | 66 | 11
Aspartate aminotransferase increased (Investigations) | 33 | 2
Alanine aminotransferase increased (Investigations) | 28 | 4
Weight increased (Investigations) | 18 | 3
Weight decreased (Investigations) | 15 | 12
Neutrophil count decreased (Investigations) | 6 | 9
Headache (Nervous system disorders) | 48 | 22
Dysgeusia (Nervous system disorders) | 28 | 12
Dizziness (Nervous system disorders) | 33 | 9
Neuropathy peripheral (Nervous system disorders) | 20 | 14
Paraesthesia (Nervous system disorders) | 13 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 8
Urinary tract infection (Infections and infestations) | 43 | 13
Upper respiratory tract infection (Infections and infestations) | 20 | 8
Rash pustular (Infections and infestations) | 15 | 2
Vision blurred (Eye disorders) | 41 | 8
Retinal detachment (Eye disorders) | 37 | 0
Dry eye (Eye disorders) | 25 | 7
Eyelid oedema (Eye disorders) | 16 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 15 | 0
Periorbital oedema (Eye disorders) | 17 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 45 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 13 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 44 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 1
Decreased appetite (Metabolism and nutrition disorders) | 55 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 28 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 6
Insomnia (Psychiatric disorders) | 32 | 12
Anxiety (Psychiatric disorders) | 21 | 6
Depression (Psychiatric disorders) | 18 | 3
Hypertension (Vascular disorders) | 46 | 4
Hot flush (Vascular disorders) | 15 | 3
Anaemia (Blood and lymphatic system disorders) | 38 | 21
Neutropenia (Blood and lymphatic system disorders) | 5 | 14
Haematuria (Renal and urinary disorders) | 15 | 1
Conjunctivitis (Eye disorders) | 12 | 3
Retinal disorder (Eye disorders) | 12 | 0
Flatulence (Gastrointestinal disorders) | 17 | 2
Influenza like illness (General disorders) | 12 | 2
Malaise (General disorders) | 13 | 4
Oedema (General disorders) | 15 | 2
Pain (General disorders) | 14 | 2
Paronychia (Infections and infestations) | 12 | 2
Blood creatinine increased (Investigations) | 14 | 2
Dehydration (Metabolism and nutrition disorders) | 13 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 1
Memory impairment (Nervous system disorders) | 3 | 6
Dysuria (Renal and urinary disorders) | 16 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 12 | 0

LIMITATIONS AND CAVEATS:
In the futility analysis based on PCD, the futility boundary was crossed, and therefore, no additional efficacy data was collected and no additional efficacy analyses were conducted. As of 01 Apr 2016, enrollment into the study were discontinued and crossover treatment was no longer permitted, any participants still receiving MEK162 were allowed to continue at the discretion of the investigator until any treatment discontinuation criterion was met and discontinued after 30-day safety follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.